CLINICAL TRIAL: NCT06664502
Title: A Phase 1/2a 2-part Study Consisting of an Open-label Multiple Ascending Dose (MAD) Safety Study in Participants With Macular Edema Following Branch Retinal Vein Occlusion (BRVO), and a Dose-finding, Double-masked, Comparative Safety, and Preliminary Efficacy Study of Intravitreal (IVT) EYE201 (Tiespectus) in Participants With Either Diabetic Macular Edema (DME) or Neovascular Age-related Macular Degeneration (NVAMD)
Brief Title: A 2-part Study Consisting of a Multiple Ascending Dose Safety Study in Participants With Macular Edema Following Branch Retinal Vein Occlusion and a Dose-finding Safety and Preliminary Efficacy Study in Participants With Either Diabetic Macular Edema or Neovascular Age-related Macular Degeneration
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EyeBiotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: EYE-TIE-201
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Macular Edema (DME); Neovascular Age-related Macular Degeneration (NVAMD); BRVO - Branch Retinal Vein Occlusion
Keywords: DME; Diabetic Macular Edema; NVAMD; Neovascular Age-related Macular Degeneration; BRVO; Branch Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Intervention Model Description: Part 1 is a multiple ascending dose (MAD) study, and patients will be enrolled sequentially in ascending order through the dose levels until the highest level is reached or until a maximum tolerated dose is reached, whichever comes first.
  Part 2 is a randomized double-masked study where patients on all arms may be enrolled in parallel.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1 MAD - Low Dose (Experimental)
  Interventions: Drug: EYE201
- Part 1 MAD - Low-Mid Dose (Experimental)
  Interventions: Drug: EYE201
- Part 1 MAD - Mid-High Dose (Experimental)
  Interventions: Drug: EYE201
- Part 1 MAD - High Dose (Experimental)
  Interventions: Drug: EYE201
- Part 2: DME naïve or experienced participants - Dose 1 (Experimental)
  Interventions: Drug: EYE201
- Part 2: DME naïve or experienced participants -Dose 2 (Experimental)
  Interventions: Drug: EYE201
- Part 2: NVAMD naïve or experienced participants - Dose 1 (Experimental)
  Interventions: Drug: EYE201
- Part 2: NVAMD naïve or experienced participants - Dose 2 (Experimental)
  Interventions: Drug: EYE201

INTERVENTIONS:
Drug: EYE201 — EYE201 solution for intravitreal administration
  Other Names: Tiespectus; MK-8748

SUMMARY:
EYE-TIE-201 is a 2-part study to investigate the safety and effectiveness of a new drug being developed called EYE201.

All participants in the study will receive a total of 3 injections of EYE201 into the study eye, spaced at 4 weeks apart.

In the first part, termed the multiple ascending dose (MAD) portion of study, the safety of EYE201 will be assessed at increasing doses in branch retinal vein occlusion (BRVO) participants. Approximately 12 participants will be entered in this part of the study.

In the second part of the study, called the dose finding part, 2 doses of EYE201 will be selected and their effectiveness will be compared. This portion of the study assesses the safety and preliminary efficacy of EYE201 in patients with diabetic macular edema (DME) or neovascular macular degeneration (NVAMD). Approximately 80 participants will be entered in this part of the study.

DETAILED DESCRIPTION:
In the multiple ascending dose (MAD) part of the study, 4 cohorts, each comprised of 3 participants, will receive IVT injections of EYE201 at one of 4 dosing levels in ascending order in an open label design. The participants will have previously untreated (naïve) BRVO and will receive EYE201.

Participants will return for safety and efficacy assessments and sample collection study visits. Participants in the following cohort will receive their first IVT injection of EYE201 once all 3 participants in the previous cohort have received their first dose of EYE201 and completed a predefined safety assessment, and a Dose Escalation Committee has confirmed the absence of dose-limiting toxicity (DLT).

Once the last participant in the MAD portion of the study has received their first dose, completed a predefined safety assessment, and the maximum tolerated dose (MTD) either has been determined or declared as not having been reached at the doses tested, 2 of the dose levels will be selected for inclusion in the Part 2 dose-finding study, based on safety and any preliminary efficacy signals observed.

The dose-finding part of the study will be randomized and masked to the participants and study site personnel (except the dose preparer and unmasked injecting physician). The study will be split according to whether the participants have treatment naïve or treatment experienced DME or NVAMD.

ELIGIBILITY:
General Key Inclusion Criteria

* Written informed consent before the first study-related activity
* Be male or female ≥ 18 years of age
* If female, have a negative serum pregnancy test at Screening and further negative urine tests immediately before each dose of study medication if the participant is a female of childbearing potential.

General Key Exclusion Criteria

* Be pregnant or breastfeeding
* Have a history of cataract surgery and/or minimally invasive glaucoma surgery in the study eye within 90 days of Screening
* Have uncontrolled blood pressure, defined as systolic ≥180 mmHg and/or diastolic ≥100 mmHg while a participant is at rest.
* Have had Yttrium-Aluminum Garnet laser capsulotomy in the study eye within 90 days of Screening
* Have had Pan-retinal Photocoagulation or focal thermal laser photocoagulation in the study eye
* Have tractional retinal detachment in the study eye
* Have uncontrolled glaucoma (defined as IOP ≥ 25 mmHg despite treatment with antiglaucoma medication) in the study eye

BRVO-specific Inclusion Criteria

Participants must:

* Be diagnosed with BRVO in the study eye
* Have a ETDRS BCVA letter score between ≤ 70 and ≥ 35 (20/40 to 20/200 Snellen equivalent) in the study eye
* Have a CST of ≥ 325 μm in the study eye on SDOCT as determined by the IRC at Screening
* Have a decrease in vision in the study eye determined by the Investigator to be primarily the result of BRVO BRVO-specific Exclusion Criteria

Participants must not:

* Have macular edema in the study eye considered to be secondary to a cause other than BRVO (e.g., DME, Irvine-Gass syndrome)
* Have active iris or angle neovascularization or neovascular glaucoma in the study eye
* Have proliferative retinopathy, central retinal vein occlusion, or hemiretinal vein occlusion

DME-specific Inclusion Criteria

Participants must:

* Have Type 1 or Type 2 diabetes mellitus and a glycated hemoglobin A1c (HbA1c) of ≤ 12%
* Have a ETDRS BCVA letter score between ≤ 70 and ≥ 35 (20/40 to 20/200 Snellen equivalent) in the study eye
* Have a CST of ≥ 325 μm in the study eye on SDOCT as determined by the IRC at Screening
* Have a decrease in vision in the study eye determined by the Investigator to be primarily the result of DME

DME-specific Exclusion Criteria

Participants must not:

* Have macular edema in the study eye considered to be secondary to a cause other than DME (eg, retinal vein occlusion, Irvine-Gass syndrome)
* Have active iris or angle neovascularization or neovascular glaucoma in the study eye
* Have high-risk proliferative diabetic retinopathy characteristics in the study eye

NVAMD-specific Inclusion Criteria

Participants must:

* Be ≥ 50 years of age
* Have a ETDRS BVCA letter score between ≤ 70 and ≥ 35 (20/40 to 20/200 Snellen equivalent) in the study eye
* Subfoveal CNV secondary to AMD, with a total lesion size (including blood, scar/atrophy & neovascularization) of ≤ 9-disc areas, of which at least 50% must be active CNV in the study eye
* Have a CST of ≥ 325 μm in the study eye on SDOCT as determined by the IRC at Screening
* Be treatment naïve with vision loss in the study eye secondary to NVAMD diagnosed within 21 days prior to the Day 1 study treatment NVAMD-specific Exclusion Criteria

Participants must not:

* Have had previous thermal subfoveal laser therapy in the study eye
* Have any subfoveal atrophy or scarring, blood over the fovea, or subfoveal fibrosis in the study eye. Additionally, no more than 25% of the total lesion size may be made up of scarring or atrophy
* Have had previous photodynamic therapy with Visudyne in the study eye
* Have diabetic retinopathy in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 12 Weeks

SECONDARY OUTCOMES:
Best- Corrected Visual Acuity | 12 Weeks

CONTACTS AND LOCATIONS:
Locations (27):
- United States (26):
  - Scottsdale, Arizona, Scottsdale, Arizona
  - Modesto, CA, Modesto, California
  - Mountain View, California, Mountain View, California
  - Sacramento, CA, Sacramento, California
  - Sacramento, California, Sacramento, California
  - Deerfield Beach, FL, Deerfield Beach, Florida
  - Lemont, IL, Lemont, Illinois
  - Hagerstown, Maryland, Hagerstown, Maryland
  - Madison, Mississippi, Madison, Mississippi
  - Bloomfield, New Jersey, Bloomfield, New Jersey
  - Asheville, NC, Asheville, North Carolina
  - Wake Forest, NC, Wake Forest, North Carolina
  - West Columbia, South Carolina, West Columbia, South Carolina
  - Germantown, Tennessee, Germantown, Tennessee
  - Knoxville, TN, Knoxville, Tennessee
  - Nashville, Tennessee, Nashville, Tennessee
  - Abilene, Texas, Abilene, Texas
  - Amarillo, Texas, Amarillo, Texas
  - Austin, Texas, Austin, Texas
  - Bellaire, Texas, Bellaire, Texas
  - Bellaire, TX, Bellaire, Texas
  - Dallas, Texas, Dallas, Texas
  - Plano, TX, Plano, Texas
  - Round Rock, TX, Round Rock, Texas
  - San Antonio, Texas, San Antonio, Texas
  - Woodlands, Texas, The Woodlands, Texas
- Arecibo, PR, Arecibo, Puerto Rico